CLINICAL TRIAL: NCT01801410
Title: Induction of Labour in Pre-eclamptic Women: a Randomised Trial Comparing the Foley Balloon Catheter With Oral Misoprostol
Brief Title: Induction With Foley OR Misoprostol (INFORM) Study
Acronym: INFORM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Gynuity Health Projects (Other); Government Dental College and Hospital, India (Other Government); Daga Memorial Women's Hospital, Nagpur, India (Other)
Responsible Party: Principal Investigator, Andrew Weeks MD MRCOG, Professor, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4001
Record Dates: First submitted 2013-02-14; First posted 2013-02-28 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Pre-eclampsia; Fetus or Newborn; Effects of Induction of Labor
Keywords: pre-eclampsia; labor induction; misoprostol; Foley catheter
MeSH Terms: conditions — Pre-Eclampsia | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): Group 2 will be induced using oral misoprostol tablets (25 mcg) every 2 hours for a maximum of 12 doses or until active labour commences. In primigravid women, if contractions have not commenced after 2 doses, the dosage may be increased to 50mcg every 2 hours. Once in labour (regular painful contractions with a cervical dilatation of at least 4cm) no more misoprostol will be used and artificial membrane rupture and/or oxytocin infusion will be used as clinically indicated. If labour has still not commenced after 24 hours, they will be deemed to have a 'failed induction' and the decision on further management will be made by the clinical team (their choice could include the use of repeat misoprostol, Foley catheter, dinoprostone, caesarean section or delay as deemed appropriate).
  Interventions: Drug: Misoprostol
- Foley Catheter (Active Comparator): Group 1 will undergo induction using a transcervical Foley catheter (silicone, size 18F with 30ml balloon) which will remain until active labour starts, the Foley catheter falls out, or 12 hours have elapsed. If the Foley catheter falls out within 12h, membranes will be ruptured and/or oxytocin infusion started. If the Foley catheter does not fall out within 12h, it will be removed at 12h and oxytocin commenced with an artificial rupture of membrane when possible. If labour has still not commenced after 24 hours, they will be deemed to have a 'failed induction' and the decision on further management will be made by the clinical team (their choice could include the use of misoprostol, repeat Foley catheter, dinoprostone, caesarean section or delay as deemed appropriate).
  Interventions: Device: Foley Catheter

INTERVENTIONS:
Device: Foley Catheter — Transcervical Foley catheter (silicone, size 18F with 30ml balloon)
  Other Names: Cervical ripening balloon, balloon catheter
  Arms: Foley Catheter
Drug: Misoprostol — 25mcg every 2 hours for maximum of 12 doses
  Other Names: Cytotec
  Arms: Misoprostol

SUMMARY:
Between 40,000 and 80,000 pregnant women die annually from pre-eclampsia and eclampsia. Magnesium sulphate and anti-hypertensive therapies can reduce the morbidity associated with pre-eclampsia. The only cure, however, comes with delivery. Prompt delivery of the baby, preferably by vaginal route, is vital in order to achieve good maternal and neonatal outcomes. Induction of labour is therefore a critical intervention in order to prevent morbidity to both mother and baby. Two low cost interventions - oral misoprostol tablets and transcervical Foley catheterization - are already used by some in low resource settings, but their relative risks and benefits are not known. These interventions could optimize the care pathway for women needing induction of labour. This is especially important in low resource settings where improvement is most needed and the potential to reduce the maternal and neonatal mortality and morbidity is the greatest. The ideal induction agent would result in a relatively short induction to delivery interval without risk to fetus and with low rates of emergency caesarean section. The induction to delivery interval is especially important in pre-eclampsia and eclampsia where the condition may deteriorate rapidly until delivery. Inductions with prostaglandins, including misoprostol, are sometimes associated with uterine hyperstimulation and consequent fetal hypoxia, whilst the effectiveness and safety of Foley catheter as an induction agent has been persistently questioned. This study will identify the risk, benefits and trade-offs in efficacy, safety, acceptability and cost of these two low cost induction methods.

DETAILED DESCRIPTION:
This is a pragmatic, open-label, randomised control trial of two methods for labour induction among women with pre-eclampsia. Women requiring delivery for preeclampsia in two hospitals in Nagpur, India will be randomised to one of two treatment groups: transcervical Foley catheter or oral misoprostol tablets.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing pregnancies with a live fetus in whom the decision has been made to induce vaginal delivery because of preeclampsia or uncontrolled hypertension. Women will be included irrespective of whether an intrapartum caesarean section on fetal grounds or would be considered or not.
* Women age ≥18 years
* Signed informed consent form

Exclusion Criteria:

* • Women with previous caesarean sections

  * Those unable to give informed consent
  * Multiple pregnancy
  * History of allergy to misoprostol
  * Ruptured membranes
  * Chorioamnionitis (by clinical diagnosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Attainment of vaginal delivery within 24 hours. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Weeks, MD FRCOG, Principal Investigator — University of Liverpool
Locations (2):
- India (2):
  - Daga Memorial Women's Hospital, Nagpur, Maharashtra
  - Government Medical College (GMC), Nagpur

REFERENCES:
- [Derived] Mundle S, Bracken H, Khedikar V, Mulik J, Faragher B, Easterling T, Leigh S, Granby P, Haycox A, Turner MA, Alfirevic Z, Winikoff B, Weeks AD. Foley catheterisation versus oral misoprostol for induction of labour in hypertensive women in India (INFORM): a multicentre, open-label, randomised controlled trial. Lancet. 2017 Aug 12;390(10095):669-680. doi: 10.1016/S0140-6736(17)31367-3. Epub 2017 Jun 28. PMID 28668289
- [Derived] Bracken H, Mundle S, Faragher B, Easterling T, Haycox A, Turner M, Alfirevic Z, Winikoff B, Weeks A. Induction of labour in pre-eclamptic women: a randomised trial comparing the Foley balloon catheter with oral misoprostol. BMC Pregnancy Childbirth. 2014 Sep 5;14:308. doi: 10.1186/1471-2393-14-308. PMID 25193157